CLINICAL TRIAL: NCT03721952
Title: Evaluating Effectiveness of a Communication Facilitator to Reduce Distress and Improve Goal Concordant Care for Critically Ill Patients and Their Families: A Randomized Trial
Brief Title: Facilitating Communication Study
Acronym: FCS2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, R. Engelberg, Research Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY00005369
Record Dates: First submitted 2018-10-16; First posted 2018-10-26 (Actual); Results first posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Chronic Disease; Neoplasm Metastasis; Lung Neoplasm; Pulmonary Disease, Chronic Obstructive; Heart Failure, Congestive; Liver Cirrhosis; Kidney Failure, Chronic; Multiple Organ Failure; Health Care Quality, Access, and Evaluation; Intensive Care Units; Palliative Care, Health Services; Palliative Care, Patient Care; Lung Diseases; Cerebrovascular Disorders; Brain Injuries
MeSH Terms: conditions — Chronic Disease; Neoplasm Metastasis; Lung Neoplasms; Pulmonary Disease, Chronic Obstructive; Heart Failure; Liver Cirrhosis; Kidney Failure, Chronic; Multiple Organ Failure; Lung Diseases; Cerebrovascular Disorders; Brain Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Facilitator-Based Intervention (Experimental): The 'Facilitator-Based Intervention' includes patient and family member subjects.
  Interventions: Behavioral: Facilitator-Based Intervention
- Usual Care (No Intervention): The 'Usual Care' arm includes patient and family member subjects.

INTERVENTIONS:
Behavioral: Facilitator-Based Intervention — Facilitators interact in person or by telephone with patients, family, and clinicians both during and following the patient's ICU stay for 3 months. In-person contacts include visits to patients' homes and/or care facilities; phone contacts include calls to patients, families and clinicians. Patients and families have access to facilitators through phone and email 5 days per week. Facilitators may attend clinic visits with patients. In addition to checking directly with patients/families during regular contacts, facilitators also access the electronic health record to ensure they have accurate information about appointments and treatment plans and to document key points for the clinical team. Facilitators encourage referral to inpatient or outpatient palliative care services when needs are identified.
  Other Names: Communication Facilitator
  Arms: Facilitator-Based Intervention

SUMMARY:
This study is a randomized clinical trial of an intervention to improve outcomes for patients and their family by using ICU nurse facilitators to support, model, and teach communication strategies that enable patients and their families to secure care in line with patients' goals of care over an illness trajectory, beginning in the ICU and continuing to care in the community.

DETAILED DESCRIPTION:
The impact of critical illness is increasing due to an aging population as well as advances in effectiveness and availability of critical care. Critically ill patients and their families suffer a high burden of symptoms of depression, anxiety, and post-traumatic stress due, in part, to fragmented medical care that is often poorly aligned with their goals. Fragmented care includes numerous transitions for patients and families across clinicians and across settings, starting in the intensive care unit (ICU) and extending to acute care, skilled nursing facilities, or home. As illness progresses, patients and families struggle to navigate the spectrum of goals of care, to match their values and goals with treatments, to communicate their goals to their clinicians, and to make difficult medical decisions without letting unmet emotional needs interfere. Poor communication exacerbated by these transitions compounds an already stressful experience, causing distress to patients and their families. Taken together, these issues lead to ineffective communication during and after the ICU which can often result in high intensity "default" care that may be unwanted.

Using a randomized trial, this project aims to evaluate an innovative model of care in which ICU nurse facilitators support, model, and teach communication strategies that enable patients and families to secure care in line with their goals over an illness trajectory, beginning in the ICU and continuing into the community. Facilitators use communication skills, attachment theory, and mediation to improve: 1) patients' and families' self-efficacy to communicate with clinicians within and across settings; 2) patients' and families' outcome expectation that communication with clinicians can improve their care; and 3) patients' and families' behavioral capability through skill building to resolve barriers to effective communication and mediate conflict. Facilitators work with seriously ill patients and their families beginning with a critical care unit stay and following them over the course of three months.

The intervention's effectiveness will be measured with patient- and family-centered outcomes at 1-, 3-, and 6-months post-randomization. The primary outcome is family members' burden of symptoms of depression over the 6 months. The investigators also evaluate whether the intervention improves the value of healthcare by reducing healthcare costs while improving patient and family outcomes. Finally, investigators use qualitative methods to explore implementation factors (intervention, settings, individuals, processes) associated with improved implementation outcomes (acceptability, fidelity, penetration) to inform dissemination of this type of intervention to support patients and their families. This study aims to address key knowledge gaps while evaluating a methodologically rigorous intervention to improve outcomes for patients with serious illness and their families across the trajectory of care and the spectrum of goals of care.

ELIGIBILITY:
Inclusion Criteria:

* PATIENTS. Eligible patients 18 years of age or older, English-speaking, with a chronic life-limiting illness suggesting a median survival of approximately 2 years or a severe acute illness with a risk of hospital mortality of at least 15%. Chronic life-limiting illnesses include: cancer with a poor prognosis (e.g. metastatic cancer); chronic pulmonary disease (e.g. COPD, restrictive lung disease); coronary artery disease (CAD); congestive heart failure (CHF); peripheral vascular disease (PVD); severe liver disease (e.g. cirrhosis); diabetes with end-organ damage; renal failure (e.g. ESRD); and dementia. Acute illness criteria include a SOFA, APACHE or trauma severity score predicting a 15% or greater risk of hospital mortality. Acute illnesses and conditions also include: age >=80 years; acute respiratory distress syndrome (ARDS) with P/F ratio <=300; subarachnoid hemorrhage (SAH) Fisher grade 3/4 with Glasgow coma score (GCS) <=12; spontaneous hemorrhage (ICH, IPH, EDH, SDH) with GCS <=12; stroke or cardiovascular accident (CVA) with GCS <=12; decompressive/crash craniotomy (bone flap) with GCS <=12; traumatic brain injury (TBI) or diffuse axonal injury (DAI) based on MRI ~day 10; or anoxic brain injury due to cardiac arrest >48 hours. All potential participants screened for facility with English and absence of significant cognitive impairment (prior to their current hospitalization) that would limit their ability to complete survey instruments.
* FAMILY. Eligible family subjects18 years of age or older, English-speaking, and identified as someone involved in patient's medical care or decision-making. Eligible family may include any of the following: legal guardians, durable power of attorney for healthcare, spouses, adult children, parents, siblings, domestic partners, other relatives, and friends.
* CLINICIAN AND ADMINISTRATOR INTERVIEW SUBJECTS. Eligible clinicians and administrators 18 years of age or older, English-speaking, employed at a participating hospital and have a familiarity with the study and the intervention.

Exclusion Criteria:

* PATIENTS. We will exclude patients with an anticipated ICU stay of less than 2 days, as assessed by the critical care attending physician or his/her designee. We will exclude patients who have been in the ICU for more than 14 days.
* PATIENTS AND FAMILY. Reasons for exclusion for patient and family member subject groups include: legal or risk management concerns (as determined by the attending physician or via hospital record designation); psychological illness or morbidity; and physical or mental limitations preventing ability to complete questionnaires.
* CLINICIAN AND ADMINISTRATOR INTERVIEW SUBJECTS. n/a

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 977 (Actual)
Dates: Start 2019-04-17 (Actual); Primary Completion 2023-10-26 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruth A Engelberg, PhD, Principal Investigator — University of Washington
Locations (3):
- United States (3):
  - UW Medicine - Harborview Medical Center, Seattle, Washington
  - University of Washington Medical Center - Northwest, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients and family were screened and recruited from April 2019 to March 2023. Potential subjects received introductory calls from the research coordinator to assess interest and eligibility. Enrollees completed baseline surveys and were randomized. Patients and family were approached for interviews between March 2020 and December 2022. Clinicians and administrators were recruited between January 2021 and January 2023.
Pre-assignment Details: 2823 patients and family were assessed for eligibility. 1806 were excluded; main reasons included: family or legal next of kin unavailable, and patient status improved/transferred from ICU. 568 declined participation; main reason given was the family member feeling overwhelmed. 505 family subjects were enrolled, representing 449 enrolled patients.
Groups:
- Usual Care/CONTROL: Patient: Received Usual Care and/or Attention Control; patient subjects did not complete surveys
- Facilitator-Based INTERVENTION: Patient: Received 3-Month Communication Facilitator Intervention; patient subjects did not complete surveys
- Usual Care/CONTROL: Family: Received Usual Care and/or Attention Control; family member subjects completed follow-up outcome surveys at 1-3-6 months after randomization
- Facilitator-Based INTERVENTION: Family: Received 3-Month Communication Facilitator Intervention; family member subjects completed follow-up outcome surveys at 1-3-6 months after randomization
- Clinician & Administrator Interviewees: Subjects participated in qualitative interviews designed to evaluate the intervention
Period: Overall Study
Arm/Group | Usual Care/CONTROL: Patient | Facilitator-Based INTERVENTION: Patient | Usual Care/CONTROL: Family | Facilitator-Based INTERVENTION: Family | Clinician & Administrator Interviewees
Started | 224 | 225 | 241 | 264 | 23
Completed Survey at 1-Month | 0 | 0 | 160 | 206 | 0
Completed Survey at 3-Months | 0 | 0 | 157 | 189 | 0
Completed Survey at 6-Months | 0 | 0 | 146 | 199 | 0
Completed Qualitative Interview | 0 | 0 | 1 | 21 | 23
Completed | 223 | 224 | 199 | 236 | 23
Not Completed | 1 | 1 | 42 | 28 | 0
Not completed — Lost to Follow-up | 0 | 0 | 2 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 40 | 28 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care/CONTROL: Patient | Facilitator-Based INTERVENTION: Patient | Usual Care/CONTROL: Family | Facilitator-Based INTERVENTION: Family | Clinician & Administrator Interviewees | Total
Number analyzed (Participants) | 224 | 225 | 241 | 264 | 23 | 977
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 58 [41 to 68] | 57 [40 to 70] | 53 [42 to 63] | 55 [43 to 64] | 39.5 [33.5 to 44.5] | 55 [41 to 66]
Age, Customized [Count of Participants; unit: Participants]
  <= 18 years | 1 | 0 | 0 | 0 | 0 | 1
  Between 18 and 65 years | 146 | 146 | 179 | 197 | 15 | 683
  >= 65 years | 77 | 79 | 54 | 63 | 1 | 274
  Unknown or Not Reported | 0 | 0 | 8 | 4 | 7 | 19
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 78 | 102 | 175 | 183 | 18 | 556
  Male | 146 | 123 | 65 | 81 | 5 | 420
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 18 | 21 | 23 | 0 | 75
  Not Hispanic or Latino | 199 | 190 | 215 | 234 | 23 | 861
  Unknown or Not Reported | 12 | 17 | 5 | 7 | 0 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 6 | 9 | 7 | 0 | 27
  Asian | 8 | 4 | 5 | 7 | 2 | 26
  Native Hawaiian or Other Pacific Islander | 3 | 2 | 4 | 2 | 0 | 11
  Black or African American | 8 | 14 | 7 | 16 | 0 | 45
  White | 186 | 180 | 190 | 205 | 19 | 780
  More than one race | 5 | 4 | 22 | 24 | 2 | 57
  Unknown or Not Reported | 9 | 15 | 4 | 3 | 0 | 31
Region of Enrollment [Number; unit: participants]
  United States | 224 | 225 | 241 | 264 | 23 | 977
Hospital Site [Count of Participants; unit: Participants]
  County Hospital | 167 | 165 | 181 | 198 | 8 | 719
  University Hospital | 45 | 46 | 47 | 51 | 11 | 200
  Community Hospital | 12 | 14 | 13 | 15 | 0 | 54
  More than One Hospital Location | 0 | 0 | 0 | 0 | 4 | 4
Diagnoses, Patients [Count of Participants; unit: Participants] — Collected from EHR. Eligibility diagnoses during the ICU stay; categorized as Chronic Condition (e.g. Dartmouth Atlas) or Acute Conditions. Counts are not mutually exclusive and participants may have more than one categorical diagnosis. Population: Measure Analysis Population Description: These data were not collected for family members ("Usual Care/CONTROL: Family" & "Facilitator-Based INTERVENTION: Family" or "Clinician & Administrator Interviewees" subjects. Patients can have more than one condition so the number will not sum to the number of participants analyzed.
  Participants
    Chronic-Cancer: number analyzed (Participants) | 224 | 225 | 0 | 0 | 0 | 449
    Chronic-Cancer | 25 | 20 | 0 | 0 | 0 | 45
    Chronic-COPD (chronic obstructive pulmonary disease): number analyzed (Participants) | 224 | 225 | 0 | 0 | 0 | 449
    Chronic-COPD (chronic obstructive pulmonary disease) | 33 | 26 | 0 | 0 | 0 | 59
    Chronic-CAD (coronary artery disease): number analyzed (Participants) | 224 | 225 | 0 | 0 | 0 | 449
    Chronic-CAD (coronary artery disease) | 38 | 34 | 0 | 0 | 0 | 72
    Chronic-CHF (congestive heart failure): number analyzed (Participants) | 224 | 225 | 0 | 0 | 0 | 449
    Chronic-CHF (congestive heart failure) | 55 | 53 | 0 | 0 | 0 | 108
    Chronic-PVD (peripheral vascular disease): number analyzed (Participants) | 224 | 225 | 0 | 0 | 0 | 449
    Chronic-PVD (peripheral vascular disease) | 26 | 12 | 0 | 0 | 0 | 38
    Chronic-Liver Disease: number analyzed (Participants) | 224 | 225 | 0 | 0 | 0 | 449
    Chronic-Liver Disease | 25 | 19 | 0 | 0 | 0 | 44
    Chronic-Diabetes: number analyzed (Participants) | 224 | 225 | 0 | 0 | 0 | 449
    Chronic-Diabetes | 17 | 22 | 0 | 0 | 0 | 39
    Chronic-Renal Failure: number analyzed (Participants) | 224 | 225 | 0 | 0 | 0 | 449
    Chronic-Renal Failure | 39 | 32 | 0 | 0 | 0 | 71
    Chronic-Dementia: number analyzed (Participants) | 224 | 225 | 0 | 0 | 0 | 449
    Chronic-Dementia | 8 | 15 | 0 | 0 | 0 | 23
    Chronic-Had 3+ Diagnoses: number analyzed (Participants) | 224 | 225 | 0 | 0 | 0 | 449
    Chronic-Had 3+ Diagnoses | 69 | 62 | 0 | 0 | 0 | 131
    Acute-ARDS (acute respiratory distress syndrome): number analyzed (Participants) | 224 | 225 | 0 | 0 | 0 | 449
    Acute-ARDS (acute respiratory distress syndrome) | 45 | 56 | 0 | 0 | 0 | 101
    Acute-On ECMO/ECLS (extracorporeal life support): number analyzed (Participants) | 224 | 225 | 0 | 0 | 0 | 449
    Acute-On ECMO/ECLS (extracorporeal life support) | 5 | 0 | 0 | 0 | 0 | 5
    Acute-TBI (traumatic brain injury): number analyzed (Participants) | 224 | 225 | 0 | 0 | 0 | 449
    Acute-TBI (traumatic brain injury) | 27 | 40 | 0 | 0 | 0 | 67
    Acute-Vascular/non-TBI (non-traumatic brain injury): number analyzed (Participants) | 224 | 225 | 0 | 0 | 0 | 449
    Acute-Vascular/non-TBI (non-traumatic brain injury) | 73 | 65 | 0 | 0 | 0 | 138
    Acute-Respiratory Failure: number analyzed (Participants) | 224 | 225 | 0 | 0 | 0 | 449
    Acute-Respiratory Failure | 177 | 174 | 0 | 0 | 0 | 351
    Acute-New spinal cord injury (SCI) with Quadriplegia: number analyzed (Participants) | 224 | 225 | 0 | 0 | 0 | 449
    Acute-New spinal cord injury (SCI) with Quadriplegia | 3 | 3 | 0 | 0 | 0 | 6
    Acute-ICU Admission with COVID-19: number analyzed (Participants) | 224 | 225 | 0 | 0 | 0 | 449
    Acute-ICU Admission with COVID-19 | 28 | 28 | 0 | 0 | 0 | 56
APACHE II Score, Patients [Median (Inter-Quartile Range); unit: APACHE II Severity of Disease Score] — Acute Physiology and Chronic Health Evaluation (APACHE II) Severity of Disease Score collected within 24-48 hours of ICU admission (where available).APACHE II gives an integer score from 0 to 71 that computed using several physiological measurements and age; higher scores correspond to more severe disease. Population: These data were not collected for family members or clinician/administrator interview subjects.
  APACHE II Severity of Disease Score
    number analyzed (Participants) | 224 | 225 | 0 | 0 | 0 | 449
    (all) | 25 [20 to 30] | 24 [19 to 30] |  |  |  | 25 [20 to 30]
Type of Insurance, Patients [Count of Participants; unit: Participants] — Population: These data were not collected for family members or clinician/administrator interview subjects.
  Participants
    number analyzed (Participants) | 224 | 225 | 0 | 0 | 0 | 449
    Private/commercial | 71 | 61 |  |  |  | 132
    Medicare | 138 | 150 |  |  |  | 288
    Military | 8 | 7 |  |  |  | 15
    Other | 6 | 6 |  |  |  | 12
    Unknown | 1 | 1 |  |  |  | 2
Relationship, Family [Count of Participants; unit: Participants] — Relationship of participating family member to the patient, self-report via survey item. Population: These data only apply to family member subjects.
  Participants
    number analyzed (Participants) | 0 | 0 | 241 | 264 | 0 | 505
    Spouse/Partner |  |  | 80 | 88 |  | 168
    Child |  |  | 62 | 71 |  | 133
    Sibling |  |  | 32 | 32 |  | 64
    Parent |  |  | 50 | 58 |  | 108
    Other relative |  |  | 10 | 8 |  | 18
    Friend |  |  | 5 | 3 |  | 8
    Other relationship |  |  | 2 | 4 |  | 6
Education Level, Family [Count of Participants; unit: Participants] — Highest completed education level of participating family member, self-report via survey item. Population: These data were only collected from family member subjects.
  Participants
    number analyzed (Participants) | 0 | 0 | 241 | 264 | 0 | 505
    8th grade or less |  |  | 1 | 0 |  | 1
    Some high school |  |  | 7 | 6 |  | 13
    High school diploma/GED |  |  | 29 | 29 |  | 58
    Trade school or some college |  |  | 103 | 121 |  | 224
    4-year college degree |  |  | 55 | 52 |  | 107
    Some graduate school |  |  | 9 | 11 |  | 20
    Graduate degree |  |  | 37 | 45 |  | 82
Employment Status, Family [Count of Participants; unit: Participants] — Employment status of participating family member, self-report via survey item. Population: These data were only collected from family member subjects.
  Participants
    number analyzed (Participants) | 0 | 0 | 241 | 264 | 0 | 505
    Full-time |  |  | 105 | 133 |  | 238
    Part-time |  |  | 27 | 23 |  | 50
    Unemployed |  |  | 20 | 18 |  | 38
    Disabled |  |  | 20 | 12 |  | 32
    Retired |  |  | 50 | 56 |  | 106
    Other |  |  | 15 | 17 |  | 32
    Unknown, not reported |  |  | 4 | 5 |  | 9
Financial Situation, Family [Count of Participants; unit: Participants] — Financial situation of participating family member, self-report via survey item. Population: These data were only collected from family member subjects.
  Participants
    number analyzed (Participants) | 0 | 0 | 241 | 264 | 0 | 505
    Enough money for special things |  |  | 107 | 119 |  | 226
    Enough money to pay bills but little for extra things |  |  | 71 | 81 |  | 152
    Enough money as a result of cutting back |  |  | 37 | 44 |  | 81
    Difficulty paying bills no matter what |  |  | 21 | 14 |  | 35
    Unknown, not reported |  |  | 5 | 6 |  | 11
Health Status, Family [Count of Participants; unit: Participants] — Health status of participating family member, self-report via Short Form Health Survey (SF-1) item. Population: These data were only collected from family member subjects.
  Participants
    number analyzed (Participants) | 0 | 0 | 241 | 264 | 0 | 505
    Excellent |  |  | 31 | 26 |  | 57
    Very Good |  |  | 93 | 107 |  | 200
    Good |  |  | 83 | 91 |  | 174
    Fair |  |  | 27 | 35 |  | 62
    Poor |  |  | 6 | 4 |  | 10
    Unknown, not reported |  |  | 1 | 1 |  | 2
Depression Symptoms, Family (HADS-D) [Mean (Standard Deviation); unit: scores on a scale] — Family member symptoms of depression and anxiety assessed with Hospital Anxiety and Depression Scale (HADS); reliable and valid 14-item, 2-domain (anxiety and depression) tool used to assess symptoms of psychological distress; 7 items evaluate anxiety and 7 evaluate depression; each item is scored on a 4-point scale (ranging from 0-3) with scores for each subscale (anxiety and depression) ranging from 0-21, with higher scores indicating greater symptoms of psychological distress. Population: These measures were only collected from family subjects. Two respondents missing data.
  scores on a scale
    number analyzed (Participants) | 0 | 0 | 240 | 263 | 0 | 503
    (all) |  |  | 7.2 (4.6) | 7.2 (4.2) |  | 7.2 (4.4)
Anxiety Symptoms, Family (HADS-A) [Mean (Standard Deviation); unit: scores on a scale] — Family member symptoms of depression and anxiety assessed with Hospital Anxiety and Depression Scale (HADS); reliable and valid 14-item, 2-domain (anxiety and depression) tool used to assess symptoms of psychological distress; 7 items evaluate anxiety and 7 evaluate depression; each item is scored on a 4-point scale (ranging from 0-3) with scores for each subscale (anxiety and depression) ranging from 0-21, with higher scores indicating greater symptoms of psychological distress. Population: These measures were only collected from family subjects. Two respondents missing data.
  scores on a scale
    number analyzed (Participants) | 0 | 0 | 240 | 263 | 0 | 503
    (all) |  |  | 10.4 (4.8) | 10.5 (4.7) |  | 10.4 (4.7)
Quality of Family Experience - Relationship with Healthcare Providers [Mean (Standard Deviation); unit: scores on a scale] — Family member measure of experience of patients with serious illness; QUAL-E (Fam) is a validated instrument to measure of quality of life at the end of life; four domains are measured, including, relationship with healthcare providers (4 items), completion (3 items), and preparation (4 items).
  These data report on the "Relationship with Healthcare Providers" subscale domain items: told what to expect, involved in decision-making, kept informed, and concerns responded to. Ratings are on a scale of 1-5, with higher score indicating 'better relationship'. Population: These measures were only collected from family subjects. Eight respondents are missing data.
  scores on a scale
    number analyzed (Participants) | 0 | 0 | 238 | 259 | 0 | 497
    (all) |  |  | 4.03 (0.81) | 4.02 (0.89) |  | 4.03 (0.85)
Quality of Family Experience - Sense of Completion [Mean (Standard Deviation); unit: scores on a scale] — Family member measure of experience of patients with serious illness; QUAL-E (Fam) is a validated instrument to measure of quality of life at the end of life; four domains are measured, including, relationship with healthcare providers (4 items), completion (3 items), and preparation (4 items).
  These data report on the "Sense of Completion" subscale domain items: able to make a positive difference, able to have meaningful interaction, and able to say important things to patient. Ratings are on a scale of 1-5, with higher score indicating 'better sense of completion'. Population: These measures were only collected from family subjects. Ten respondents are missing data.
  scores on a scale
    number analyzed (Participants) | 0 | 0 | 236 | 259 | 0 | 495
    (all) |  |  | 3.38 (1.28) | 3.32 (1.27) |  | 3.35 (1.27)
Quality of Family Experience - Preparation Issues [Mean (Standard Deviation); unit: scores on a scale] — Family member measure of experience of patients with serious illness; QUAL-E (Fam) is a validated instrument to measure of quality of life at the end of life; four domains are measured, including, relationship with healthcare providers (4 items), completion (3 items), and preparation (4 items)
  These data report on the "Preparation" subscale domain items: feeling financial strain, feeling emotionally prepared for future, feeling at peace, feeling at peace patient's care. Ratings are on a scale of 1-5, with higher score indicating 'better preparation'. Population: These measures were only collected from family subjects. Two respondents are missing data.
  scores on a scale
    number analyzed (Participants) | 0 | 0 | 241 | 262 | 0 | 503
    (all) |  |  | 13.5 (3.0) | 13.3 (3.3) |  | 13.4 (3.2)
Goal-Concordant Care, Family Assessment [Count of Participants; unit: Participants] — Family report on concordance between the care patients want and the care they are receiving; measured with two 'forced choice' items: 1) patient preference (would the patient prefer a course of treatment focused on extending life as much as possible, even if it means having more pain and discomfort, or would the patient want a plan of care focused on relieving pain and discomfort as much as possible, even if that means not living as long?); and 2) perception of current treatment using the same two options. If the answers on the two items matched, they were considered "concordant". Population: These measures were only collected from family subjects. Twelve respondents are missing data.
  Participants
    number analyzed (Participants) | 0 | 0 | 232 | 261 | 0 | 493
    (all) |  |  | 123 | 136 |  | 259
Perceived Competence, FAMILY [Median (Inter-Quartile Range); unit: units on a scale] — The Perceived Competence Scale (PCS) is a 4-item questionnaire assessing participants' feelings of competence. Items can be worded differently for different target behaviors. Responses range from "Not at all true" (1) to "Very True" (7); higher score on the latent variable would indicate greater competence. We will evaluate this mediator cross-sectionally. Population: This measure was only collected from family subjects.
  units on a scale
    I feel confident in my ability to get the care for my family member that he/she wants.: number analyzed (Participants) | 0 | 0 | 221 | 244 | 0 | 465
    I feel confident in my ability to get the care for my family member that he/she wants. |  |  | 6 [5 to 7] | 6 [4 to 7] |  | 6 [4 to 7]
    I am capable of getting the care for my family member that he/she wants.: number analyzed (Participants) | 0 | 0 | 222 | 243 | 0 | 465
    I am capable of getting the care for my family member that he/she wants. |  |  | 6 [4 to 7] | 6 [4 to 7] |  | 6 [4 to 7]
    I am able to get the care for my family member that he/she wants.: number analyzed (Participants) | 0 | 0 | 221 | 244 | 0 | 465
    I am able to get the care for my family member that he/she wants. |  |  | 6 [4 to 7] | 6 [4 to 7] |  | 6 [4 to 7]
    I feel able to meet the challenge of getting the care for my family member that he/she wants.: number analyzed (Participants) | 0 | 0 | 223 | 242 | 0 | 465
    I feel able to meet the challenge of getting the care for my family member that he/she wants. |  |  | 6 [4 to 7] | 6 [4 to 7] |  | 6 [4 to 7]

OUTCOME MEASURES:

1. Primary Outcome: Depression Symptoms, Family (HADS-D)
Description: Family member symptoms of depression and anxiety assessed with the Hospital Anxiety and Depression Scale (HADS). The HADS is a reliable and valid 14-item, 2-domain (anxiety and depression) tool used to assess symptoms of psychological distress. Seven items evaluate anxiety and seven evaluate depression. Each item is scored on a 4-point scale (ranging from 0-3.
  For each of three follow-up points (1-month, 3-month, and 6-month), the response variable was the sum of 7 items measuring depression, weighted for the number of items with valid responses. The sum could range from 0 to 21, with higher values indicating greater depression (i.e., worse outcome),
Time Frame: 1-month, 3-month, and 6-month values for the outcome, using a linear mixed-effects model that evaluates the effects of the intervention, time point, and the intervention-time interaction on the outcome after adjustment for the baseline value
Population: Family members with answers to at least half (4 of 7) of the HADS depression items at baseline and also with answers to at least half of the HADS depression items at one or more of the three follow-up points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care/CONTROL: Family | Facilitator-Based INTERVENTION: Family
Number analyzed (Participants) | 191 | 235
score on a scale
  at 1-month: number analyzed (Participants) | 160 | 206
  at 1-month | 6.4 (4.4) | 6.5 (4.3)
  at 3-months: number analyzed (Participants) | 157 | 189
  at 3-months | 6.3 (4.3) | 5.9 (4.1)
  at 6-months: number analyzed (Participants) | 145 | 199
  at 6-months | 5.9 (4.1) | 5.9 (4.5)
Statistical Analysis 1: Comparison: Facilitator-Based INTERVENTION: Family; Superior outcome for Group2 (Facilitator-based INTERVENTION: Family); Test type: Superiority; p = 0.688, Mixed Models Analysis; Linear mixed-effects: 1-, 3-, 6-mo outcomes, intervention & time predictors. Primary analysis: avg control-intervention effect over 3 time points; Avg. Intervention Effect (CON--INT) = 0.130, 95% CI 2-sided [-0.505 to 0.764], Standard Error of Mean 0.323 — Additional estimation information: Positive sign of estimate defined as lower average depression score & negative sign of estimate defined as higher average depression score, over 3 follow-up points for the intervention group vs. the control group
Statistical Analysis 2: Comparison: Facilitator-Based INTERVENTION: Family; Test type: Superiority; p = 0.510, Mixed Models Analysis; Average Intervention effect with time interaction (control-intervention)

2. Secondary Outcome: Anxiety Symptoms, Family (HADS-A)
Description: Family member symptoms of depression and anxiety assessed with the Hospital Anxiety and Depression Scale (HADS). The HADS is a reliable and valid 14-item, 2-domain (anxiety and depression) tool used to assess symptoms of psychological distress. Seven items evaluate anxiety and seven evaluate depression. Each item is scored on a 4-point scale (ranging from 0-3. For each of three follow-up points (1-month, 3-month, and 6-month), the response variable was the sum of 7 items measuring anxiety, weighted for the number of items with valid responses. The sum could range from 0 to 21, with higher values indicating greater anxiety (i.e., worse outcome)
Time Frame: as for outcome 1
Population: Family members with answers to at least half (4 of 7) of the HADS anxiety items at baseline and also with answers to at least half of the HADS anxiety items at one or more of the three follow-up points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care/CONTROL: Family | Facilitator-Based INTERVENTION: Family
Number analyzed (Participants) | 191 | 235
score on a scale
  at 1-month: number analyzed (Participants) | 160 | 206
  at 1-month | 8.2 (4.5) | 8.4 (4.3)
  at 3-months: number analyzed (Participants) | 157 | 189
  at 3-months | 8.4 (4.8) | 8.2 (4.4)
  at 6-months: number analyzed (Participants) | 146 | 199
  at 6-months | 8.1 (4.8) | 7.9 (4.6)
Statistical Analysis 1: Comparison: Facilitator-Based INTERVENTION: Family; Superior outcome for Group2 (Facilitator-based INTERVENTION: Family); Test type: Superiority; p = 0.658, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Avg. Intervention Effect (CON--INT) = 0.143, 95% CI 2-sided [-0.491 to 0.777], Standard Error of Mean 0.323 — Additional estimation information: Positive sign of estimate defined as lower average anxiety score & negative sign of estimate defined as higher average anxiety score, over 3 follow-up points for the intervention group vs. the control group
Statistical Analysis 2: Comparison: Facilitator-Based INTERVENTION: Family; Test type: Superiority; p = 0.268, Mixed Models Analysis; Average Intervention effect with time interaction (control-intervention)

3. Secondary Outcome: Quality of Family Experience - Relationship With Healthcare Providers (QUAL-E Fam)
Description: Measure of family experience of patients with serious illness. The QUAL-E (Fam) is a validated 17-item companion instrument to the patient QUAL-E measure of quality of life at the end of life, with four subscales and two general items. This study is using 11 items from three subscales: Relationship with Health Care Provider, Completion, and Preparation subscales. For each of three follow-up points (1-month, 3-month, and 6-month), the response variable was the mean of the valid responses to QUAL-E (Fam) items #5, 6, 7, and 8. The mean could range from 1 to 5, with higher values indicating higher quality of relationship (i.e., better outcome).
Time Frame: as for outcome 1
Population: Family members with answers to at least half (2 of 4) of QUAL-E (Fam) items #5, 6, 7, and 8 at baseline and also with answers to at least half of those items at one or more of the three follow-up points; higher score indicates higher quality of relationship.
Measure: Mean (Standard Deviation); unit: score on a scale, mean value of 4 items
Arm/Group | Usual Care/CONTROL: Family | Facilitator-Based INTERVENTION: Family
Number analyzed (Participants) | 184 | 217
score on a scale, mean value of 4 items
  at 1-month: number analyzed (Participants) | 162 | 204
  at 1-month | 3.94 (0.85) | 4.10 (0.77)
  at 3-months: number analyzed (Participants) | 108 | 132
  at 3-months | 3.51 (1.16) | 3.87 (0.97)
  at 6-months: number analyzed (Participants) | 84 | 127
  at 6-months | 3.54 (1.13) | 3.64 (1.11)
Statistical Analysis 1: Comparison: Facilitator-Based INTERVENTION: Family; Superior outcome for Group 2 (Facilitator-based INTERVENTION: Family); Test type: Superiority; p = 0.010, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Avg. Intervention Effect (CON--INT) = -0.200, 95% CI 2-sided [-0.353 to -0.048], Standard Error of Mean 0.077 — Additional information: Positive sign of estimate defined as lower average quality-of-relationship score & negative sign of estimate defined as higher average quality-of-relationship score over 3 follow-up points for intervention vs control groups
Statistical Analysis 2: Comparison: Facilitator-Based INTERVENTION: Family; Test type: Superiority; p = 0.175, Mixed Models Analysis; Average Intervention effect with time interaction (control-intervention)

4. Secondary Outcome: Quality of Family Experience - Sense of Completion (QUAL-E Fam)
Description: Measure of family experience of patients with serious illness. The QUAL-E (Fam) is a validated 17-item companion instrument to the patient QUAL-E measure of quality of life at the end of life, with four subscales and two general items. This study is using 11 items from three subscales: Relationship with Health Care Provider, Completion, and Preparation subscales. For each of three follow-up points (1-month, 3-month, and 6-month), the response variable was the mean of the valid responses to QUAL-E (Fam) items #9, 10, and 11. The mean could range from 1 to 5, with higher values indicating higher sense of completion (i.e., better outcome).
Time Frame: as for outcome 1
Population: Family members with answers to at least half (2 of 3) of QUAL-E (Fam) items #9, 10, and 11 at baseline and also with answers to at least half of those items at one or more of the three follow-up points; higher score indicates higher sense of completion.
Measure: Mean (Standard Deviation); unit: score on a scale, mean value of 3 items
Arm/Group | Usual Care/CONTROL: Family | Facilitator-Based INTERVENTION: Family
Number analyzed (Participants) | 184 | 217
score on a scale, mean value of 3 items
  at 1-month: number analyzed (Participants) | 162 | 203
  at 1-month | 3.68 (1.16) | 3.75 (1.02)
  at 3-months: number analyzed (Participants) | 111 | 137
  at 3-months | 3.98 (0.98) | 3.94 (1.03)
  at 6-months: number analyzed (Participants) | 91 | 136
  at 6-months | 4.05 (0.93) | 4.01 (1.00)
Statistical Analysis 1: Comparison: Facilitator-Based INTERVENTION: Family; Superior outcome for Group 2 (Facilitator-based INTERVENTION: Family); Test type: Superiority; p = 0.817, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Avg. Intervention Effect (CON--INT) = -0.021, 95% CI 2-sided [-0.203 to 0.160], Standard Error of Mean 0.092 — Additional information: Positive sign of estimate defined as lower average quality-of-relationship score & negative sign of estimate defined as higher average quality-of-relationship score, over 3 follow-up points for intervention vs control group
Statistical Analysis 2: Comparison: Facilitator-Based INTERVENTION: Family; Test type: Superiority; p = 0.949, Mixed Models Analysis; Average Intervention effect with time interaction (control-intervention)

5. Secondary Outcome: Quality of Family Experience - Preparation Issues (QUAL-E Fam)
Description: Measure of family experience of patients with serious illness. The QUAL-E (Fam) is a validated 17-item companion instrument to the patient QUAL-E measure of quality of life at the end of life, with four subscales and two general items. This study is using 11 items from three subscales: Relationship with Health Care Provider, Completion, and Preparation subscales. For each of three follow-up points (1-month, 3-month, and 6-month), the response variable was the sum of valid responses to QUAL-E (Fam) items #12, 13, 14, and 15, weighted for the number of items with valid responses. The sum could range from 4 to 20, with higher values indicating greater preparation (i.e., better outcome).
Time Frame: as for outcome 1
Population: Family members with answers to at least half (2 of 4) of QUAL-E (Fam) items #12, 13, 14, and 15 at baseline and also with answers to at least half of those items at one or more of the three follow-up points; higher score indicates higher preparation.
Measure: Mean (Standard Deviation); unit: score on a scale, sum of items
Arm/Group | Usual Care/CONTROL: Family | Facilitator-Based INTERVENTION: Family
Number analyzed (Participants) | 190 | 222
score on a scale, sum of items
  at 1-month: number analyzed (Participants) | 163 | 207
  at 1-month | 13.5 (3.2) | 13.9 (3.2)
  at 3-months: number analyzed (Participants) | 112 | 137
  at 3-months | 13.3 (3.2) | 14.0 (3.2)
  at 6-months: number analyzed (Participants) | 92 | 137
  at 6-months | 13.6 (3.4) | 14.0 (3.2)
Statistical Analysis 1: Comparison: Facilitator-Based INTERVENTION: Family; Superior outcome for Group 2 (Facilitator-based INTERVENTION: Family); Test type: Superiority; p = 0.060, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Avg. Intervention Effect (CON--INT) = -0.450, 95% CI 2-sided [-0.919 to 0.020], Standard Error of Mean 0.239 — Additional information: Positive sign of estimate defined as lower average preparation score & negative sign of estimate defined as higher average preparation score, over 3 follow-up points for intervention vs control group
Statistical Analysis 2: Comparison: Facilitator-Based INTERVENTION: Family; Test type: Superiority; p = 0.701, Mixed Models Analysis; Average Intervention effect with time interaction (control-intervention)

6. Secondary Outcome: Goal-Concordant Care, Family Assessment
Description: Concordance between the care patients want and the care they receive is measured with two questions from the SUPPORT study. The first defines preference (care focused on extending life even with more pain and discomfort vs. care focused on relieving pain and discomfort even with not living as long.) The second assesses perception of current treatment using the same options. The outcome is a dichotomous variable of whether preference matches care received. For each of three follow-up points (1-month, 3-month, and 6-month), the response variable was coded 1 if the respondent's perception of the focus of care the patient received (comfort vs. life extension) matched their perception of the patient's preferred focus of care; and 0 if the perceived focus of care received did not match the perceived patient's care preference. If the response to either item was "don't know," the outcome was coded 0. The higher value indicated goal-concordant care (the better outcome).
Time Frame: as for outcome 1
Population: Family members who - at baseline - provided valid responses to both component items or who said "don't know" to either item; and who also at one or more of the follow-up points - provided valid responses to both component items or who said "don't know" to either item.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care/CONTROL: Family | Facilitator-Based INTERVENTION: Family
Number analyzed (Participants) | 182 | 219
score on a scale
  at 1-month: number analyzed (Participants) | 160 | 200
  at 1-month | 0.57 (0.497) | 0.63 (0.484)
  at 3-months: number analyzed (Participants) | 108 | 137
  at 3-months | 0.57 (0.497) | 0.65 (0.479)
  at 6-months: number analyzed (Participants) | 92 | 131
  at 6-months | 0.59 (0.495) | 0.64 (0.481)
Statistical Analysis 1: Comparison: Facilitator-Based INTERVENTION: Family; Superior outcome for Group 2 (Facilitator-based INTERVENTION: Family); Test type: Superiority; p = 0.053, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Avg. Intervention Effect (CON--INT) = -0.393, 95% CI 2-sided [-0.791 to 0.005] — Additional estimation information: Positive sign of estimate defined as lower average goal-concordant care & negative sign of estimate defined as higher average goal-concordant care, over 3 follow-up points for intervention group vs. control group
Statistical Analysis 2: Comparison: Facilitator-Based INTERVENTION: Family; Test type: Superiority; p = 0.039, Mixed Models Analysis; Average Intervention effect with time interaction (control-intervention)

7. Secondary Outcome: Impact of Event, Family Assessment (IES-6)
Description: The Impact of Event Scale-6 (IES-6), derived from the IES-R, uses six self-report items to assess subjective distress caused by a traumatic event. Items are rated on a 5-point scale ranging from 0 ("not at all") to 4 ("extremely"). For each of three follow-up points (1-month, 3-month, and 6-month), the response variable was the sum of 6 items measuring the traumatic impact of events, weighted for the number of items with valid responses. The sum could range from 0 to 24, with higher values indicating greater traumatic impact (i.e., worse outcome)
Time Frame: 1-month, 3-month, and 6-month values for the outcome, using a linear mixed-effects model that evaluates the effects of the intervention, time point, and the intervention-time interaction on the outcome
Population: Family members with answers to at least half (3 of 6) of the IES items at one or more of the three follow-up points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care/CONTROL: Family | Facilitator-Based INTERVENTION: Family
Number analyzed (Participants) | 189 | 234
score on a scale
  at 1-month: number analyzed (Participants) | 155 | 202
  at 1-month | 11 (6) | 9.4 (5.9)
  at 3-months: number analyzed (Participants) | 150 | 184
  at 3-months | 9 (6) | 8.9 (6.4)
  at 6-months: number analyzed (Participants) | 145 | 192
  at 6-months | 9 (6) | 8.1 (6.0)
Statistical Analysis 1: Comparison: Facilitator-Based INTERVENTION: Family; Superior outcome for Group2 (Facilitator-based INTERVENTION: Family); Test type: Superiority; p = 0.239, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Avg. Intervention Effect (CON--INT) = 0.636, 95% CI 2-sided [-0.425 to 1.700]
Statistical Analysis 2: Comparison: Facilitator-Based INTERVENTION: Family; Test type: Superiority; p = 0.170, Mixed Models Analysis; Average Intervention effect with time interaction (control-intervention)

8. Secondary Outcome: Healthcare Utilization: Hospital Readmission - Patient
Description: Documentation in the patient's electronic health record of hospital readmission within 30 days after discharge from the index hospitalization: 0=no readmission, 1=one or more readmissions; missing if index hospitalization still ongoing at the end of the 183-day follow-up period, patient death during index hospitalization, or randomization occurred after index hospitalization discharge. Valid outcomes could be either 0 or 1, with higher value indicating a worse outcome.
Time Frame: within 30 days after discharge from the index hospitalization
Population: Patients whose index hospitalization had ended before the end of the 183-day follow-up period, who did not die during the index hospitalization, and who were randomized before index hospitalization discharge.
Measure: Mean (Standard Deviation); unit: score on a scale (0,1)
Groups:
- Usual Care/CONTROL: Patient: Received Usual Care and/or Attention Control
- Facilitator-Based INTERVENTION: Patient: Received 3-Month Communication Facilitator Intervention
Arm/Group | Usual Care/CONTROL: Patient | Facilitator-Based INTERVENTION: Patient
Number analyzed (Participants) | 144 | 157
score on a scale (0,1) | 0.10 (0.31) | 0.19 (0.39)
Statistical Analysis 1: Comparison: Facilitator-Based INTERVENTION: Patient; Superior outcome for Group2 (Patient-Intervention); Test type: Superiority; p = 0.029, Regression, Linear; Linear regression of outcome on group (0=control, 1=interv), adjusted for hospital, w robust standard error estimate using bias correction 1/(1-h)^2; Slope = 0.089, 95% CI 2-sided [0.009 to 0.169], Standard Error of Mean 0.041 — Additional estimation information: Positive sign of estimate defined as higher proportion of readmissions & negative sign of estimate defined as lower proportion of readmissions, for the intervention group vs. the control group

9. Secondary Outcome: Healthcare Utilization: Hospital Free Days, 30 Days - Patient
Description: Number of full days on which the patient was alive and not in the hospital between the randomization date and 29 days after the randomization date. Values could range from 0 to 30, with higher value indicating a better outcome; missing if randomization occurred after index hospitalization discharge.
Time Frame: 30 days after randomization
Population: Patients who were randomized before index hospitalization discharge.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Usual Care/CONTROL: Patient | Facilitator-Based INTERVENTION: Patient
Number analyzed (Participants) | 220 | 223
days | 5.65 (8.45) | 6.78 (8.74)
Statistical Analysis 1: Comparison: Facilitator-Based INTERVENTION: Patient; Superior outcome for Group2 (Patient-Intervention); Test type: Superiority; p = 0.183, Regression, Linear; [statistical method as in outcome 8, analysis 1]; Slope = 1.078, 95% CI 2-sided [-0.511 to 2.666], Standard Error of Mean 0.808 — Additional estimation information: Positive sign of estimate defined as higher number of hospital free days & negative sign of estimate defined as lower number of hospital free days, for the intervention group vs. the control group

10. Secondary Outcome: Healthcare Utilization: Hospital Free Days, 91 Days - Patient
Description: Number of full days on which the patient was alive and not in the hospital between the randomization date and 90 days after the randomization date. Values could range from 0 to 91, with higher value indicating a better outcome; missing if randomization occurred after index hospitalization discharge.
Time Frame: 91 days after randomization
Population: Patients who were randomized before index hospitalization discharge.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Usual Care/CONTROL: Patient | Facilitator-Based INTERVENTION: Patient
Number analyzed (Participants) | 220 | 223
days | 39.63 (32.95) | 41.43 (33.29)
Statistical Analysis 1: Comparison: Facilitator-Based INTERVENTION: Patient; Superior outcome for Group2 (Patient-Intervention); Test type: Superiority; p = 0.593, Regression, Linear; [statistical method as in outcome 8, analysis 1]; Slope = 1.687, 95% CI 2-sided [-4.518 to 7.892], Standard Error of Mean 3.157 — [estimate comment as in outcome 9, analysis 1]

11. Secondary Outcome: Healthcare Utilization: Hospital Free Days, 183 Days - Patient
Description: Number of full days on which the patient was alive and not in the hospital between the randomization date and 182 days after the randomization date. Values could range from 0 to 183, with higher value indicating a better outcome; missing if randomization occurred after index hospitalization discharge.
Time Frame: 183 days after randomization
Population: Patients who were randomized before index hospitalization discharge.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Usual Care/CONTROL: Patient | Facilitator-Based INTERVENTION: Patient
Number analyzed (Participants) | 220 | 223
days | 93.66 (74.03) | 98.13 (72.55)
Statistical Analysis 1: Comparison: Facilitator-Based INTERVENTION: Patient; Superior outcome for Group2 (Patient-Intervention); Test type: Superiority; p = 0.533, Regression, Linear; [statistical method as in outcome 8, analysis 1]; Slope = 4.365, 95% CI 2-sided [-9.367 to 18.097], Standard Error of Mean 6.987 — [estimate comment as in outcome 9, analysis 1]

12. Secondary Outcome: Healthcare Utilization: ICU Free Days, 30 Days - Patient
Description: Number of full days on which the patient was alive and not in an ICU between the randomization date and 29 days after the randomization date. Values could range from 0 to 30, with higher value indicating a better outcome; missing if randomization occurred after index hospitalization discharge.
Time Frame: 30 days after randomization
Population: Patients who were randomized before index hospitalization discharge.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Usual Care/CONTROL: Patient | Facilitator-Based INTERVENTION: Patient
Number analyzed (Participants) | 220 | 223
days | 18.54 (11.90) | 19.62 (10.59)
Statistical Analysis 1: Comparison: Facilitator-Based INTERVENTION: Patient; Superior outcome for Group2 (Patient-Intervention); Test type: Superiority; p = 0.318, Regression, Linear; [statistical method as in outcome 8, analysis 1]; Slope = 1.070, 95% CI 2-sided [-1.032 to 3.173], Standard Error of Mean 1.070 — Additional estimation information: Positive sign of estimate defined as higher number of ICU free days & negative sign of estimate defined as lower number of ICU free days, for the intervention group vs. the control group

13. Secondary Outcome: Healthcare Utilization: ICU Free Days, 91 Days - Patient
Description: Number of full days on which the patient was alive and not in an ICU between the randomization date and 90 days after the randomization date. Values could range from 0 to 91, with higher value indicating a better outcome; missing if randomization occurred after index hospitalization discharge.
Time Frame: 91 days after randomization
Population: Patients who were randomized before index hospitalization discharge.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Usual Care/CONTROL: Patient | Facilitator-Based INTERVENTION: Patient
Number analyzed (Participants) | 220 | 223
days | 58.20 (38.20) | 62.32 (35.32)
Statistical Analysis 1: Comparison: Facilitator-Based INTERVENTION: Patient; Superior outcome for Group2 (Patient-Intervention); Test type: Superiority; p = 0.241, Regression, Linear; [statistical method as in outcome 8, analysis 1]; Slope = 4.117, 95% CI 2-sided [-2.773 to 11.007], Standard Error of Mean 3.506 — [estimate comment as in outcome 12, analysis 1]

14. Secondary Outcome: Healthcare Utilization: ICU Free Days, 183 Days - Patient
Description: Number of full days on which the patient was alive and not in an ICU between the randomization date and 182 days after the randomization date. Values could range from 0 to 183, with higher value indicating a better outcome; missing if randomization occurred after index hospitalization discharge.
Time Frame: 183 days after randomization
Population: Patients who were randomized before index hospitalization discharge.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Usual Care/CONTROL: Patient | Facilitator-Based INTERVENTION: Patient
Number analyzed (Participants) | 220 | 223
days | 113.96 (80.66) | 122.15 (76.32)
Statistical Analysis 1: Comparison: Facilitator-Based INTERVENTION: Patient; Superior outcome for Group2 (Patient-Intervention); Test type: Superiority; p = 0.273, Regression, Linear; [statistical method as in outcome 8, analysis 1]; Slope = 8.195, 95% CI 2-sided [-6.479 to 22.868], Standard Error of Mean 7.466 — [estimate comment as in outcome 12, analysis 1]

15. Secondary Outcome: Healthcare Costs, Discharge - Patient
Description: Total hospitalization costs from date of randomization to index hospitalization discharge. Costs ranged from $1,631.73 to $1,299,781.53, with higher value indicating a worse outcome; missing if the patient was randomized after discharge from the index hospitalization.
Time Frame: Randomization to discharge from index hospitalization, up to 183 days
Population: Patients who were randomized before index hospitalization discharge.
Measure: Mean (Standard Deviation); unit: USDollar (inflation-adjusted total cost)
Arm/Group | Usual Care/CONTROL: Patient | Facilitator-Based INTERVENTION: Patient
Number analyzed (Participants) | 220 | 223
USDollar (inflation-adjusted total cost) | 124,358.13 (144,023.29) | 129,058.54 (156,741.01)
Statistical Analysis 1: Comparison: Facilitator-Based INTERVENTION: Patient; Superior outcome for Group2 (Patient-Intervention); Test type: Superiority; p = 0.710, other type of regression; Regression [gamma family, link function g(u)=u-0.9], outcome on random group (0=control, 1=intervention), adjusted for hospital, robust SEs; Slope = -0.0000009, 95% CI 2-sided [-0.0000057 to 0.0000039], Standard Error of Mean 0.00000248

16. Secondary Outcome: Healthcare Costs, 30 Days - Patient
Description: Total hospitalization costs for the 30-day period beginning with the date of randomization, adjusted to their value in December 2023 based on the Consumer Price Index for Medical Care. Values ranged from $1,631.73 to $585,386.34, with higher values indicating worse outcomes; missing if the patient was randomized after index hospitalization discharge.
Time Frame: Randomization to 30 days after randomization
Population: Patients who were randomized before index hospitalization discharge.
Measure: Mean (Standard Deviation); unit: USDollar (inflation-adjusted total cost)
Arm/Group | Usual Care/CONTROL: Patient | Facilitator-Based INTERVENTION: Patient
Number analyzed (Participants) | 220 | 223
USDollar (inflation-adjusted total cost) | 103,731.28 (86,239.93) | 99,087.38 (82,595.41)
Statistical Analysis 1: Comparison: Facilitator-Based INTERVENTION: Patient; Superior outcome for Group2 (Patient-Intervention); Test type: Superiority; p = 0.599, other type of regression; Regression [inverse Gaussian family, link function g(u)=u-0.9], outcome on random group (0=control,1=intervention), adjusted for hospital, robust SEs; Slope = 0.00000113, 95% CI 2-sided [-0.0000030 to 0.0000053], Standard Error of Mean 0.00000215

17. Other Pre Specified Outcome: Perceived Competence Scale (PCS), 1 Month - Family
Description: The Perceived Competence Scale (PCS) is a 4-item questionnaire assessing participants' feelings of competence. Items can be worded differently for different target behaviors. Responses range from "Not at all true" (1) to "Very True" (7); higher score on the latent variable would indicate greater competence. We will evaluate this mediator cross-sectionally.
Time Frame: Assessed on 1-month questionnaires
Population: Perceived Competence Scale, 4 items collected by self-report via survey item at each assessment point. These data were only collected from family member subjects. Unit of Measure is self-assessed competence (1 [not at all true] through 3 [somewhat true] to 7 [very true]). PCS was not asked in after-death questionnaires. Number analyzed only reflects valid responses (not skipped or missing).
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Usual Care/CONTROL: Family | Facilitator-Based INTERVENTION: Family
Number analyzed (Participants) | 241 | 264
score on a scale
  I feel confident in my ability to get the care for my family member that he/she wants.: number analyzed (Participants) | 106 | 154
  I feel confident in my ability to get the care for my family member that he/she wants. | 5 [4 to 7] | 6 [4 to 7]
  I am capable of getting the care for my family member that he/she wants.: number analyzed (Participants) | 106 | 155
  I am capable of getting the care for my family member that he/she wants. | 5 [4 to 7] | 6 [4 to 7]
  I am able to get the care for my family member that he/she wants.: number analyzed (Participants) | 105 | 155
  I am able to get the care for my family member that he/she wants. | 5 [4 to 6] | 5 [4 to 7]
  I feel able to meet the challenge of getting the care for my family member that he/she wants.: number analyzed (Participants) | 105 | 153
  I feel able to meet the challenge of getting the care for my family member that he/she wants. | 5 [4 to 7] | 5 [4 to 7]

18. Other Pre Specified Outcome: Perceived Competence Scale (PCS), 3 Months - Family
Description: as for outcome 17
Time Frame: Assessed on 3-month questionnaires
Population: as for outcome 17
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Usual Care/CONTROL: Family | Facilitator-Based INTERVENTION: Family
Number analyzed (Participants) | 241 | 264
score on a scale
  I feel confident in my ability to get the care for my family member that he/she wants.: number analyzed (Participants) | 95 | 122
  I feel confident in my ability to get the care for my family member that he/she wants. | 5 [4 to 7] | 6 [4 to 7]
  I am capable of getting the care for my family member that he/she wants.: number analyzed (Participants) | 95 | 121
  I am capable of getting the care for my family member that he/she wants. | 5 [4 to 6] | 6 [4 to 7]
  I am able to get the care for my family member that he/she wants.: number analyzed (Participants) | 96 | 121
  I am able to get the care for my family member that he/she wants. | 5 [4 to 6] | 6 [4 to 6]
  I feel able to meet the challenge of getting the care for my family member that he/she wants.: number analyzed (Participants) | 96 | 121
  I feel able to meet the challenge of getting the care for my family member that he/she wants. | 5 [4 to 6] | 6 [4 to 7]

19. Other Pre Specified Outcome: Perceived Competence Scale (PCS), 6 Months - Family
Description: as for outcome 17
Time Frame: Assessed on 6-month questionnaires
Population: as for outcome 17
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Usual Care/CONTROL: Family | Facilitator-Based INTERVENTION: Family
Number analyzed (Participants) | 241 | 264
score on a scale
  I feel confident in my ability to get the care for my family member that he/she wants.: number analyzed (Participants) | 84 | 132
  I feel confident in my ability to get the care for my family member that he/she wants. | 6 [4 to 7] | 6 [4 to 6.75]
  I am capable of getting the care for my family member that he/she wants.: number analyzed (Participants) | 84 | 131
  I am capable of getting the care for my family member that he/she wants. | 6 [4 to 7] | 6 [4 to 7]
  I am able to get the care for my family member that he/she wants.: number analyzed (Participants) | 85 | 130
  I am able to get the care for my family member that he/she wants. | 5 [4 to 6.5] | 5 [4 to 6]
  I feel able to meet the challenge of getting the care for my family member that he/she wants.: number analyzed (Participants) | 85 | 131
  I feel able to meet the challenge of getting the care for my family member that he/she wants. | 5 [4 to 7] | 5 [4 to 7]

20. Other Pre Specified Outcome: Measure of Acceptability of Intervention - Family in the Intervention Group
Description: The "Acceptability of Intervention Measure" (AIM) is a 4 item measure with proven reliability, validity and responsiveness to change. It is designed to assess participants' perception of the intervention in which they participated as agreeable ("meets my approval"), palatable ("appealing to me") or satisfactory ("like it", "welcome it"). Response options include "completely disagree", "disagree", "neither agree nor disagree", "agree" and "completely agree". These items were asked of the intervention participants at the conclusion of the 3-month intervention phase.
Time Frame: Assessed on 3-month questionnaires
Population: These questionnaire items were only asked of the family subjects in the intervention arm. Reporting valid responses on the 3-month questionnaire distributed at the end of the intervention period.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Usual Care/CONTROL: Family | Facilitator-Based INTERVENTION: Family
Number analyzed (Participants) | 0 | 264
score on a scale
  The facilitator intervention meets my approval.: number analyzed (Participants) | 0 | 182
  The facilitator intervention meets my approval. |  | 5 [5 to 5]
  The facilitator intervention is appealing to me.: number analyzed (Participants) | 0 | 182
  The facilitator intervention is appealing to me. |  | 5 [4.25 to 5]
  I like the facilitator intervention.: number analyzed (Participants) | 0 | 180
  I like the facilitator intervention. |  | 5 [5 to 5]
  I welcome the facilitator intervention.: number analyzed (Participants) | 0 | 179
  I welcome the facilitator intervention. |  | 5 [5 to 5]

21. Other Pre Specified Outcome: Key Implementation Factors
Description: Qualitative interviews after individual participation. Interviews will be guided by the Consolidated Framework for Implementation Research (CFIR) to explore the factors associated with implementation, including aspects of the intervention, inner and outer settings, individuals, and processes of care. Individual constructs within these domains were chosen to fit this specific intervention and context.
Time Frame: 6-months after randomization
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Key Implementation Outcomes
Description: Qualitative interviews after individual participation. Interviews will also explore three key implementation outcomes (acceptability, fidelity, penetration) that will guide future dissemination of the intervention.
Time Frame: 6-months after randomization
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Enrollment/Randomization though 6-month study duration
Arm/Group | Usual Care/CONTROL: Patient | Facilitator-Based INTERVENTION: Patient | Usual Care/CONTROL: Family | Facilitator-Based INTERVENTION: Family | Clinician & Administrator Interviewees
All-Cause Mortality (participants affected / at risk) | 111/224 | 94/225 | 0/241 | 0/264 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/224 | 0/225 | 0/241 | 0/264 | 0/23
Other Adverse Events (participants affected / at risk) | 0/224 | 0/225 | 0/241 | 0/264 | 0/23

LIMITATIONS AND CAVEATS:
This study took place in one region of the US and may not generalize to other regions. There may be selection bias among those family members and patients who were willing to participate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-10): https://cdn.clinicaltrials.gov/large-docs/52/NCT03721952/Prot_SAP_000.pdf